CLINICAL TRIAL: NCT06843616
Title: A PILOT TRIAL of a DISPOSABLE INTRACEREBRAL ASPIRATION ENDOSCOPE for the TREATMENT of INTRACEREBRAL HEMATOMA（FAST-HET）
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: MicroPort NeuroTech Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NeuroFlash-2024-01-CIP-00
Record Dates: First submitted 2025-01-08; First posted 2025-02-25 (Actual); Last update posted 2025-02-25 (Actual); Status verified 2025-02

CONDITIONS: Intracerebral Hemorrhage
MeSH Terms: conditions — Cerebral Hemorrhage | interventions — Endoscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Endoscopic surgery (Experimental): Using a disposable intracerebral aspiration endoscope to remove the intracerebral hematoma
  Interventions: Procedure: Endoscopic surgery

INTERVENTIONS:
Procedure: Endoscopic surgery — Using a disposable intracerebral aspiration endoscope to remove the intracerebral hematoma

SUMMARY:
This clinical trial is a prospective, open-label, single-arm clinical trial. According to the inclusion and exclusion criteria specified in the trial protocol, no fewer than 16 subjects with cerebral hemorrhage will be enrolled in 1 to 2 clinical centers. Considering the learning period required for doctor to become proficient in using the device, the first three cases at each research center are considered as the lead-in period cases and will not be included in the primary analysis dataset. During the surgery, a disposable intracerebral aspiration endoscope will be used to remove the intracerebral hematoma. Follow-ups will be conducted at discharge/Day 7 (±1 day), postoperative 1 month (±7 days), and postoperative 3 months (±15 days). Recording various indicators to evaluate the safety and effectiveness of the disposable intracerebral aspiration endoscope in treating intracerebral hematoma.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 and ≤ 80 years old;
2. Spontaneous intracerebral hemorrhage;
3. Hemorrhage located in the supratentorial subcortical or basal ganglia region;
4. Hematoma volume ≥ 30ml and ≤ 80ml;
5. Able to undergo surgery within 72 hours after onset;
6. GCS score of 5 to 14;
7. The subject themselves and/or their authorized representative can understand the purpose of the study, agree to participate, and sign the informed consent form.

Exclusion Criteria:

1. History of intracerebral hemorrhage within the past year;
2. Traumatic intracerebral hemorrhage;
3. Multiple intracerebral hemorrhages;

   Note: Hemorrhage in the supratentorial subcortical or basal ganglia region that extends into the ventricles is not considered multiple hemorrhages and can be included.
4. Known or suspected intracerebral hemorrhage caused by tumors, aneurysms, vascular malformations, hemorrhagic transformation of ischemic stroke, cerebral venous thrombosis, etc.;
5. Formation of brain herniation;
6. Severe neurological or psychiatric disorders before onset (such as epilepsy, Alzheimer's disease, Parkinson's disease, schizophrenia, depression, etc.);
7. mRS score ≥ 3 before onset;
8. Use of anticoagulants or antiplatelet drugs within 14 days before onset, or the need for long-term use of anticoagulants or antiplatelet drugs, or other factors causing coagulation dysfunction;
9. Platelet count less than 100 × 10^3/μL or international normalized ratio (INR) greater than 1.4;
10. Active bleeding present, such as gastrointestinal bleeding, respiratory bleeding, or subcutaneous hematoma;
11. Uncontrolled hypertension that cannot be managed with medication (systolic blood pressure > 220 mmHg or diastolic blood pressure > 120 mmHg after medication upon admission);
12. Severe systemic diseases that cannot tolerate surgery, such as severe liver or kidney dysfunction;
13. Women of childbearing age who are pregnant or breastfeeding;
14. Currently participating in any drug or device research, or planning to participate in other drug or device clinical trials;
15. Life expectancy ≤ 1 year;
16. Other situations where the researcher deems the subject unsuitable for the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2025-02-06 (Actual); Primary Completion 2025-08-31 (Estimated); Study Completion 2025-10-31 (Estimated)

PRIMARY OUTCOMES:
Intracerebral hematoma clearance rate | Day 0（within 24 hours after procedure）
  Perform a brain CT scan within 24 hours after surgery, comparing it with the baseline CT, and calculating the proportion of hematoma volume reduction.

SECONDARY OUTCOMES:
Hospitalization duration | During the days at hospital(up to 105 days)
Intensive Care Unit(ICU) duration | During the days at Intensive Care Unit(ICU)(up to 105 days)
The proportion of subjects with an mRS score of ≤3 at 3 months after surgery | 3 months after surgery(±15days)
The incidence of rebleeding at the surgical site within 7 days after surgery or before discharge. | 7 days (±1day) after surgery or before discharge.
The incidence of reoperation due to rebleeding at the surgical site during the follow-up period. | 3 months after surgery(±15days)
All-cause mortality | 3 months after surgery(±15days)
Device-related SAE | 3 months after surgery(±15days)

CONTACTS AND LOCATIONS:
Locations (1):
- Affiliated Hospital of Guizhou Medical University, Guiyang, Guizhou, China

IPD SHARING:
Plan to Share IPD: No